CLINICAL TRIAL: NCT00743483
Title: An Open Label, Exploratory Study on the Effect of rhBSSL on the Fat Absorption in Patients With Cystic Fibrosis and Pancreatic Insufficiency
Brief Title: Efficacy of Bucelipase Alfa (BSSL) in Patients With Cystic Fibrosis and Pancreatic Insufficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BVT.BSSL-002; 2007-004063-21 (EudraCT Number)
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Cystic Fibrosis; Exocrine Pancreatic Insufficiency
Keywords: cystic fibrosis; pancreatic insufficiency; bucelipase alfa; bile salt stimulating lipase; BSSL; coefficient of fat absorption
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rhBSSL (Experimental): 170 mg rhBSSL three times daily for 5 to 6 consecutive days
  Interventions: Drug: rhBSSL

INTERVENTIONS:
Drug: rhBSSL — oral suspension, 170 mg BSSL, 3 times daily for 5-6 days
  Other Names: BSSL, Bucelipase alfa, rhBSSL

SUMMARY:
The purpose of this study is to evaluate the efficacy in patients with cystic fibrosis and pancreatic insufficiency following treatment with BSSL

DETAILED DESCRIPTION:
In this open study, patients will enter a baseline period of 6 days where the pancreatic enzyme therapy will be discontinued and a standard diet given. After the baseline period, patients will enter a treatment period of 6 days where a fixed dose of BSSL will be administered. The primary efficacy measurements will be made by collecting stool during the last three days of each period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cystic fibrosis and pancreatic insufficiency who are able to refrain from their ongoing pancreatic enzyme treatment for a period of 7 days and are able to produce stools >= 5 times per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Isal, MD, PhD, Study Director — Swedish Orphan Biovitrum; Janneke Langendonk, MD, PhD, Principal Investigator — Erasmus Medical Center, Rotterdam, Netherlands
Locations (4):
- Erasmus Medical Center, Rotterdam, Netherlands
- Poland (3):
  - Specjalistyczny Zespól Opieki Zdrowotnej nad Matka i Dzieckiem w Gdansku, Gdansk
  - Uniwersytet Medyczny im. K. Marcinkowskiego, Poznan
  - Oddzialu Terenowego Instytutu, Gruzlicy i Chorob Pluc w Rabce-Zdroju, Rabka-Zdrój

RESULTS

PARTICIPANT FLOW:
Groups:
- rhBSSL: Oral suspension, 170 mg rhBSSL, 3 times daily for 5-6 days
Period: Baseline Period
Arm/Group | rhBSSL
Started | 15
Completed | 14
Not Completed | 1
Not completed — Physician Decision | 1
Period: Treatment Period
Arm/Group | rhBSSL
Started | 14
Completed | 13
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- BSSL: Bucelipase alfa (INN): oral suspension, 170 mg BSSL, 3 times daily for 5-6 days
Arm/Group | BSSL
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.4 (10.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Poland | 12
  Netherlands | 3

OUTCOME MEASURES:

1. Primary Outcome: The Absolute Difference Between Baseline and Treatment Coefficient of Fat Absorption (CFA)
Description: The absolute difference between baseline and treatment CFA, i.e. the change from the baseline level.
  CFA was calculated as follows 100 x ((fat consumed - fat excreted)/fat consumed).
  Fat consumed was determined from the weight of fat of the dietary intake during a 72 hour period during the final 3 days of the baseline and treatment period.
  Fat excreted was determined from stool collected during the 72-hour periods and analyzed for fat using the Van de Kamer method.
  The unit of CFA is %
Time Frame: Final 3 days of baseline and treatment period
Population: Per protocol
Measure: Mean (Standard Deviation); unit: % CFA
Groups:
- rhBSSL: oral suspension, 170 mg, 3 times daily for 5-6 days
Arm/Group | rhBSSL
Number analyzed (Participants) | 9
% CFA | 6.9 (15.56)
Statistical Analysis 1: Comparison: rhBSSL; Test type: Superiority or Other; p = 0.2179, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Treatment period (5-6 days)
Description: Only treatment emergent events (events that started post-rhBSSL administration) is presented
Groups:
- BSSL: Oral suspension, 170 mg, 3 times daily for 5-6 days
Arm/Group | BSSL
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 6/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BSSL (N=14)
Cystic Fibrosis Exacerbation (Congenital, familial and genetic disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BSSL (N=14)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Viral Infection (Infections and infestations) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other